CLINICAL TRIAL: NCT05990751
Title: Multi-modular Chimeric Antigen Receptor Targeting GD2 in Neuroblastoma
Acronym: MAGNETO
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL\142424
Record Dates: First submitted 2023-08-05; First posted 2023-08-14 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Neuroblastoma
Keywords: neuroblastoma; CAR T cells
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GD2 CAR T cells (Experimental): Treatment with GD2 CAR T cells
  Interventions: Biological: GD2 CAR T cells

INTERVENTIONS:
Biological: GD2 CAR T cells — The GD2 CAR T cells target GD2 positive cells. The cells also express transgenes that aim to increase their resistance within the tumour microenvironment.

SUMMARY:
MAGNETO is a single-centre, non-randomised, open label Phase I clinical trial of an Advanced Therapy Investigational Medicinal Product (ATIMP) in children and teenagers aged 1-16 years with relapsed or refractory neuroblastoma.

The study will assess the feasibility of generating the ATIMP (GD2 CAR T cells) and the safety of administering the ATIMP in patients with relapsed or refractory neuroblastoma.

DETAILED DESCRIPTION:
MAGNETO is a single-centre, non-randomised, open label Phase I clinical trial of an Advanced Therapy Investigational Medicinal Product (ATIMP) in children and teenagers aged 1-16 years with neuroblastoma.

The ATIMP for this study (GD2 CAR T cells) are autologous T cells, modified to express GD2 CAR (targeting GD2 on the neuroblastoma cells) and additional transgenes aiming to confer resistance to inhibition in the tumour microenvironment and to support CAR T cell function and persistence.

Patients will undergo an unstimulated leucapheresis for the generation of the ATIMP which will take approximately 15 days to generate.

Patients will receive lymphodepleting (LD) chemotherapy with fludarabine 30 mg/m2 administered over 4 days (Day -6 to Day -3) and cyclophosphamide 500 mg/m2 administered over 2 days (Day -4 and Day-3).

Patients will be treated at one of three dose levels following LD chemotherapy as described above.

The study will evaluate the feasibility of generating the ATIMP, the safety of administering ATIMP, the tolerability of the ATIMP and how effectively the CAR T cells engraft, expand and persist following administration in patients with neuroblastoma.

Following infusion of the CAR T cells, patients will be monitored for between 2-4 weeks as an inpatient. Following discharge, patients will enter the interventional follow up phase and be followed up for 1 year. Patients will be seen at 6 weeks post infusion then 3 monthly until 1 year post CAR T cells infusion.

If patients relapse within the first-year post CAR T cell infusion, they will come off the interventional follow up and will be followed up annually until 15 years after the CAR T infusion.

After completing the 1-year interventional phase of the study, all patients, irrespective of whether they progressed or responded to treatment, will enter long term follow up until 15 years post CAR T infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 1 and ≤ 16 years.
2. Tissue diagnosis of neuroblastoma. If sufficient biopsy material is available, GD2 expression on the tumour will be confirmed. As GD2 is consistently expressed in neuroblastoma demonstration of GD2 is not mandated.
3. Disease which has relapsed after or is refractory to at least one line of salvage combination chemotherapy.
4. Measurable disease by cross sectional imaging or evaluable disease by uptake on 123I-MIBG scan. Patients with only bone marrow detectable disease (bone marrow aspirate or trephine) are NOT eligible for the study.
5. At least 3 weeks or 5 half-lives, whichever is shorter, after treatment with agents on other early phase clinical trial.
6. Performance status: Karnofsky (age ≥ 10 years) or Lansky (age < 10) score ≥ 50%. Patients who are unable to walk because of paralysis, but who are able to sit upright unassisted in a wheelchair, will be considered ambulatory for the purpose of assessing performance score.
7. Creatinine ≤1.5 ULN for age, if higher, an estimated (calculated) creatinine clearance must be ≥ 60 ml/min/1.73 m2.
8. Absolute lymphocyte count ≥ 0.25 x 10^9/L.
9. For post-pubertal subjects agreement to have a pregnancy test, use adequate contraception (if applicable).
10. Written informed consent.

Exclusion Criteria:

1. Patients with only bone marrow detectable disease in the absence of measurable disease by cross sectional imaging or evaluable disease by uptake on 123I-MIBG scan.
2. Patients with active, inoperative CNS disease including leptomeningeal disease.
3. Active hepatitis B, C or HIV infection.
4. Inability to tolerate leukapheresis.
5. Clinically significant systemic illness or medical condition (e.g., significant cardiac, pulmonary, hepatic or other organ dysfunction), that in the judgement of the investigator is likely to interfere with assessment of safety or efficacy of the investigational regimen and its requirements.
6. Any contraindication to lymphodepletion or to the use of Cyclophosphamide or Fludarabine as per the local SmPC.
7. Any contraindication to the use of Anticoagulant Citrate Dextrose Solution.
8. Known allergy to albumin, EDTA or DMSO.
9. Primary immunodeficiency or history of autoimmune disease (e.g., Crohn's, rheumatoid arthritis, systemic lupus) requiring systemic immunosuppression /systemic disease modifying agents within the last 2 years.
10. Prior treatment with investigational or approved gene therapy or cell therapy products.
11. Life expectancy <3 months.
12. Use of rituximab (or rituximab biosimilar) within the last 3 months prior to of GD2 CAR T cells infusion.
13. Systemic corticosteroid therapy ≥ 0.05 mg/kg dexamethasone daily (or equivalent) at time of GD2 CAR T cells infusion.
14. Post-pubertal subjects who are pregnant or breastfeeding.

Exclusion criteria for the ATIMP infusion:

1. Uncontrolled fungal, bacterial, viral, or other infection. Previously diagnosed infection for which the patient continues to receive antimicrobial therapy is permitted if responding to treatment and clinically stable at the time of scheduled GD2 CAR T cells infusion.
2. Systemic corticosteroid therapy ≥ 0.05 mg/kg dexamethasone daily (or equivalent) at time of GD2 CAR T cells infusion.
3. Use of rituximab (or rituximab biosimilar) within the last 3 months prior to GD2 CAR T cell infusion

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2041-12 (Estimated)

PRIMARY OUTCOMES:
Safety of administering the ATIMP | 28 days
  Incidence of grade 3-5 toxicity causally related to the ATIMP, particularly severe cytokine release syndrome and severe neurotoxicity.
Number of therapeutic products generated and the number of ATIMPs infused after successful manufacture | 28 days
  Feasibility of generation of the ATIMP as evaluated by the number of therapeutic products generated and the number of ATIMPs infused after successful manufacture.

SECONDARY OUTCOMES:
Objective response rate | 1 year
  Based on cross-sectional imaging and semi-quantitative assessment on 123I-MIBG after the ATIMP intravenous administration
Progression Free Survival (PFS) | 1 year
  Progression Free Survival (PFS) after the ATIMP intravenous administration
Time to Progression (TTP) | 1 year
  Time to Progression (TTP) after the ATIMP intravenous administration
Overall survival | 1 year
  Overall Survival after the ATIMP intravenous administration

CONTACTS AND LOCATIONS:
Locations (1):
- Great Ormond Street Hospital, London, United Kingdom